CLINICAL TRIAL: NCT00528931
Title: A Phase 1, Open-Label Study to Assess the Pharmacokinetics and Safety of a Single Injection of AA4500 0.58 mg in Subjects With Dupuytren's Contracture
Brief Title: A Pharmacokinetic Study of AA4500 (XIAFLEX™, Proposed Name) in Subjects With Dupuytren's Contracture
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AUX-CC-855
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Results first posted 2012-08-20 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Dupuytren's Contracture
Keywords: Assessment of AUX I and/or AUX II in human plasma
MeSH Terms: conditions — Dupuytren Contracture | interventions — Microbial Collagenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AA4500 0.58 mg (Experimental)
  Interventions: Biological: collagenase clostridium histolyticum

INTERVENTIONS:
Biological: collagenase clostridium histolyticum — Single dose of AA4500 0.58 mg into the cord
  Other Names: XIAFLEX®; AA4500

SUMMARY:
A Phase 1, open-label, single-dose pharmacokinetic study in subjects with Dupuytren's contracture conducted at one site in the United States. All subjects received a single dose of AA4500 0.58 mg, which was injected directly into the cord affecting either the metacarpophalangeal (MP) or proximal interphalangeal (PIP) joint. Pharmacokinetic blood samples were collected before dosing, at predetermined time points through the 24 hours after dosing, Day 7, and Day 30. Efficacy and safety assessments were performed up to 30 days after the AA4500 0.58 injection.

This study was designed to be part of the larger clinical program, for adult patients with Dupuytren's contracture with a palpable cord, where the data from 2 pivotal Placebo-Controlled studies (AUX-CC-857 [NCT00528606]and AUX-CC-859 [NCT00533273]) and 7 non-pivotal studies were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of Dupuytren's contracture, with a fixed flexion deformity of at least one finger, other than the thumb, that had a contracture at least 20°, but not greater than 100° for MP (80° for PIP) joints, caused by a palpable cord.
* Had a positive "table top test," defined as the inability to simultaneously place the affected finger(s) and palm flat against a table top.
* Were naive to AA4500 treatment.
* Were judged to be in good health.

Exclusion Criteria:

* Had a chronic muscular, neurological, or neuromuscular disorder that affected the hands.
* Had received treatment for Dupuytren's contracture within 90 days of the AA4500 injection to the MP or PIP selected, including surgery (fasciectomy or surgical fasciotomy), needle aponeurotomy/fasciotomy, or injection of verapamil and/or interferon on the selected primary joint within 90 days before the first dose of study drug.
* Had a known recent history of stroke, bleeding, a disease process that affected the hands, or other medical condition, which in the investigator's opinion, would make the subject unsuitable for enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Urdaneta, MD, Study Director — Endo Pharmaceuticals
Locations (1):
- Providence Clinical Research, Burbank, California, United States

REFERENCES:
- See also: XIAFLEX Prescribing Information — http://www.accessdata.fda.gov/drugsatfda_docs/label/2010/125338lbl.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- AA4500 0.58 mg: collagenase clostridium histolyticum 0.58mg injected into either the metacarpophalangeal (MP) or proximal interphalangeal (PIP) joint
Period: Overall Study
Arm/Group | AA4500 0.58 mg
Started | 16
Completed | 15
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 15
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1
  White | 14
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With AUX I and AUX II Detected in Their Blood After a Single Dose of AA4500
Description: AUX I and AUX II are the constituent protein collagenases of collagenase clostridium histolyticum (AA4500). Plasma concentrations of AUX I and AUX II were assessed through an enzymye-linked-immunoabsorbent assay (ELISA).
Time Frame: Before dosing, at predetermined time points through the 24 hours after dosing, Day 7, and Day 30
Population: Pharmacokinetic population
Measure: Number; unit: participants
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 16
participants | 0

2. Secondary Outcome: Clinical Success
Description: Clinical success defined as a reduction in contracture (ie, flexion deformity) to ≤5° of normal as measured by finger goniometry 30 days after an injection. Last observation carried forward (LOCF) after the injection was used if the status at day 30 could not be determined.
Time Frame: 30 days after treatment to the primary joint
Population: Efficacy assessment based on safety population which included all enrolled subjects who received the AA4500 injection
Measure: Number; unit: Percentage of joints
Units Other Than Participants: Joints
Groups:
- AA4500 0.58 mg: Collagenase clostridium histolyticum 0.58 mg injected into either the MP or PIP joint
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 16
Number analyzed (Joints) | 16
Percentage of joints | 75.0

3. Secondary Outcome: Clinical Improvement
Description: Clinical improvement defined as ≥50% reduction from baseline in contracture within 30 days of the injection. LOCF after the injection was used if the status at day 30 could not be determined.
Time Frame: 30 days after treatment to the primary joint
Population: Efficacy assessment based on safety population which included all enrolled subjects who received the AA4500 injection.
Measure: Number; unit: Percentage of joints
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 16
Number analyzed (Joints) | 16
Percentage of joints | 100.0

4. Secondary Outcome: Percent Change From Baseline Contracture
Description: Change from baseline in the degree of fixed-flexion contracture calculated as 100 times (baseline contracture minus last available post-injection contracture measurement) divided by baseline contracture where a positive change indicates a reduction in the degree of contracture.
Time Frame: Baseline, 30 days after treatment to the primary joint
Population: Efficacy assessment based on safety population which included all enrolled subjects who received the AA4500 injection.
Measure: Mean (Standard Deviation); unit: Percentage of contracture change
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 16
Number analyzed (Joints) | 16
Percentage of contracture change | 91.6 (16.57)

5. Secondary Outcome: Change From Baseline Range of Motion
Description: Range of motion defined as the difference between the finger extension angle and finger flexion angle expressed in degrees
Time Frame: Baseline, 30 days after treatment to the primary joint
Population: Efficacy assessment based on safety population which included all enrolled subjects who received the AA4500 injection.
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 16
Number analyzed (Joints) | 16
Degrees | 39.1 (15.38)

ADVERSE EVENTS:
Time Frame: From the time that the first dose of study drug was administered until 30 days elapsed following discontinuation of study drug administration.
Description: This study was designed to be part of the larger clinical program. For information regarding XIAFLEX-associated Serious and Non-serious Adverse events please refer to the XIAFLEX Medication Guide & XIAFLEX Prescribing Information (see links above).
Arm/Group | AA4500 0.58 mg
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 0.58 mg (N=16)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 0.58 mg (N=16)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Blood urine present (Investigations) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Injection site haemorrhage (General disorders) | 15 (15)
Injection site oedema (General disorders) | 1 (1)
Injection site pain (General disorders) | 13 (13)
Injection site swelling (General disorders) | 14 (14)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Auxilium Pharmaceuticals, Inc. agreements may vary with individual investigators but will not prohibit any investigator from publishing. Auxilium supports the publication of results from all centers of a multicenter trial but requests that reports based on single site data not preceed the primary publication of the entire clinical trial.